CLINICAL TRIAL: NCT05263960
Title: A Multicenter, Open Label, Phase I/II Clinical Study of CM350 in Patients With Advanced Solid Tumors
Brief Title: A Study of CM350 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM350-030001
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation phase in phase I (Experimental): There are 11 target dose levels in dose escalation phase.
  Interventions: Biological: CM350 group1
- Dose expansion phase in phase I (Experimental): Three or four doses will be selected for further evaluation in dose expansion phase to determine the RP2D (recommended phase 2 dose).
  Interventions: Biological: CM350 group2
- Phase II (Experimental): The efficacy of CM350 will be evaluated at RP2D (recommended phase 2 dose) for advanced GPC3-positive solid tumors.
  Interventions: Biological: CM350 group3

INTERVENTIONS:
Biological: CM350 group1 — CM350 will be administered intravenously (IV) once a week (QW) through step-up dosing until the participant discontinues study treatment, develops disease progression, initiates a new anti-tumor therapy, develops unacceptable toxicity, death, lost to follow-up, the investigator discontinue study treatment, or a female participant becomes pregnant (whichever occurs first).
  Arms: Dose escalation phase in phase I
Biological: CM350 group2 — CM350 will be administered intravenously (IV) once a week (QW) through step-up dosing until the participant discontinues study treatment, develops disease progression, initiates a new anti-tumor therapy, develops unacceptable toxicity, death, lost to follow-up, the investigator discontinue study treatment, or a female participant becomes pregnant (whichever occurs first).
  Arms: Dose expansion phase in phase I
Biological: CM350 group3 — CM350 will be administered intravenously (IV) once a week (QW). Individual subjects may continue study treatment until the participant discontinues study treatment, develops disease progression, initiates a new anti-tumor therapy, develops unacceptable toxicity, death, lost to follow-up, the investigator discontinue study treatment, or a female participant becomes pregnant (whichever occurs first).
  Arms: Phase II

SUMMARY:
This is an open label, dose escalation and expansion Phase I/II study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of CM350 in patients with advanced solid tumors.

The phase I study consists of a dose escalation phase and a dose expansion phase The safety and tolerability of CM350 and the maximum tolerated dose (MTD) (if applicable) will be evaluated in dose escalation phase.

The recommended phase 2 dose (RP2D) of CM350 will be determined in dose expansion phase.

The phase II study is to evaluate the efficacy of CM350 at the recommended phase 2 dose (RP2D) for advanced glypican-3 (GPC3)-positive solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically or cytologically confirmed advanced solid tumors that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
* hepatocellular-cancer(HCC) participants must have a Barcelona Clinic Liver Cancer (BCLC) stage of B (ineligible for liver surgery and/or other locoregional treatments, or disease progression after locoregional therapy) or stage C , or a China National Liver Cancer (CNLC) stage of IIb or III (ineligible for liver surgery and/or other locoregional treatments, or disease progression after locoregional therapy).
* HCC participants must have a Child-Pugh score of ≤7.
* Phase I dose escalation phase: participants must have evaluable lesions based on RECIST version 1.1.Phase I dose expansion phase and phase II: participants must have at least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Patients who have received any cytotoxic chemotherapy, radiotherapy, biological therapy (oncologic vaccines, cytokines, or growth factors for cancer control), or any other investigational anticancer drug treatment (defined as treatments without regulatory approval for any indication) within 28 days before the first dose of CM350.

Note: For palliative radiotherapy to non-central nervous system lesions (total radiotherapy duration ≤14 days) to improve symptoms, a minimum washout period of 7 days before the first dose is required.

* Patients who have received any immunotherapy (including but not limited to PD-1, PD-L1, anti-cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4], chimeric antigen receptor T-cell [CAR-T] therapy, etc.) within 28 days or 5 half-lives (whichever is shorter) before the first dose of CM350.
* Patients who have received targeted therapy within 28 days or 5 half-lives (whichever is shorter) before the first dose of CM350.
* Patients who have previously received any therapy targeting GPC3, including but not limited to monoclonal antibodies, peptide vaccines, CAR-T, and bispecific antibodies.
* Received chronic systemic corticosteroid therapy (daily intake of more than 10 mg prednisone or equivalent doses of other corticosteroids) or any other form of immunosuppressive treatment within 7 days before the first dose of CM350.
* Known active central nervous system metastases. Note: Participants with previously treated brain metastases that have been stable for at least 14 days before the first dose (confirmed by repeat imaging at least 4 weeks apart, with the repeat imaging conducted during the screening period) may be considered for enrollment.
* Participants with uncontrolled pleural effusion, ascites, or pericardial effusion as assessed by the investigator.
* History of other malignancies within 5 years before the first dose of CM350, excluding cured basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, or ductal carcinoma in situ of the breast.
* Presence of active infection at screening as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Dose escalation phase in phase I:Incidence of Adverse events（AEs）, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing. | Up to 5 years
  Incidence of Adverse events（AEs）, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Dose escalation phase in phase I:Dose-Limiting Toxicity (DLT). | Up to 7 days after the first target dose
  Dose-Limiting Toxicity (DLT).
Dose escalation phase in phase I:Maximum tolerated dose (MTD) (if applicable). | Up to the end of dose escalation phase (3 years)
  Maximum tolerated dose (MTD) (if applicable).
Dose expansion phase in phase I:To determine the recommended Phase 2 Dose (RP2D). | Up to 5 years
  the efficacy including objective response rate (ORR), disease control rate (DCR), etc., safety, pharmacokinetics (PK) and pharmacodynamics (PD) profile of CM350 will be assessed.
Phase II:To evaluate the efficacy of CM350 in advanced glypican-3-positive solid tumors. | Up to 5 years
  including objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (Modified Response Evaluation Criteria in Solid Tumors [mRECIST] for liver cancer and RECIST v1.1) evaluated by investigator.

SECONDARY OUTCOMES:
Phase I & Phase II: Area Under the Curve from 0 to the time of the last quantifiable concentration (AUC0-t). | Up to 5 years
  After first and multiple dosing
Phase I & Phase II: To assess the incidence of anti-drug antibody (ADA). | Up to 5 years
  To assess the incidence of anti-drug antibody (ADA)
Phase I: To evaluate the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 [Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for liver cancer and RECIST v1.1]. | Up to 5 years
  To evaluate the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 [Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for liver cancer and RECIST v1.1]
Phase I & Phase II: To evaluate the duration of response (DOR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1). | Up to 5 years
  To evaluate the duration of response (DOR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1)
Phase I & Phase II: To evaluate the disease control rate (DCR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1). | Up to 5 years
  To evaluate the disease control rate (DCR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1)
Phase I & Phase II:To evaluate the time to response (TTR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1. | Up to 5 years
  To evaluate the time to response (TTR) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1
Phase I & Phase II:To evaluate the time to progression (TTP) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1). | Up to 5 years
  To evaluate the time to progression (TTP) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1)
Phase I & Phase II:To evaluate the progression-free survival (PFS) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1). | Up to 5 years
  To evaluate the progression-free survival (PFS) per RECIST v1.1(mRECIST for liver cancer and RECIST v1.1)
Phase I & Phase II:To evaluate the overall survival (OS) | Up to 5 years
  To evaluate the overall survival (OS)
Phase I & Phase II:To assess the cytokine interleukin-2 (IL-2). | Up to 5 years
  To assess the pharmacokinetic (PD) profile of CM350.
Phase II:Incidence of Adverse events（AEs）, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing. | Up to 5 years
  Incidence of Adverse events（AEs）, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Phase I & Phase II:Area Under the Curve over a dosing interval (AUC tau). | Up to 5 years
  Area Under the Curve over a dosing interval (AUC tau).
Phase I & Phase II:Peak Plasma Concentration (Cmax). | Up to 5 years
  Peak Plasma Concentration (Cmax)
Phase I & Phase II:Time of Maximum Observed Concentration (Tmax). | Up to 5 years
  Time of Maximum Observed Concentration (Tmax)
Phase I & Phase II:Observed concentration at the end of a dosing interval (Ctrough). | Up to 5 years
  Observed concentration at the end of a dosing interval (Ctrough)
Phase I & Phase II:To assess the cytokine interleukin-6 (IL-6). | Up to 5 years
  To assess the cytokine interleukin-6 (IL-6)
Phase I & Phase II:To assess the cytokine interleukin-10 (IL-10). | Up to 5 years
  To assess the cytokine interleukin-10 (IL-10)
Phase I & Phase II:To assess the cytokine interferon-gamma(IFN-γ). | Up to 5 years
  To assess the cytokine interferon-gamma(IFN-γ)
Phase I & Phase II:To assess the cytokine tumor necrosis factor-alpha (TNF-α). | Up to 5 years
  To assess the cytokine tumor necrosis factor-alpha (TNF-α)
Phase I & Phase II: To assess the Immunophenotyping cluster of differentiation 3 positive (CD3+). | Up to 5 years
  To assess the Immunophenotyping cluster of differentiation 3 positive (CD3+).
Phase I & Phase II: To assess the Immunophenotyping cluster of differentiation 4 positive (CD4+). | Up to 5 years
  To assess the Immunophenotyping cluster of differentiation 4 positive (CD4+).
Phase I & Phase II: To assess the Immunophenotyping cluster of differentiation 8 positive (CD8+). | Up to 5 years
  To assess the Immunophenotyping cluster of differentiation 8 positive (CD8+).

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai